CLINICAL TRIAL: NCT00809835
Title: Galantamine to Enhance Cognitive Behavioral Therapy for Cocaine Abuse With Methadone Maintained Individuals
Brief Title: Galantamine to Enhance Cognitive Behavioral Therapy for Cocaine Abuse
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 0708002943; R01DA015969-13 (NIH)
Record Dates: First submitted 2008-12-16; First posted 2008-12-17 (Estimated); Results first posted 2017-06-12 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Cocaine Dependence
Keywords: Cocaine; Methadone; CBT
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Galantamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Standard Treatment As Usual (TAU) (No Intervention): Standard Treatment plus placebo for cocaine abusing or dependent methadone-maintained individuals. This consists of daily methadone visits plus one individual and one group session per week, and patients may participate in additional treatments such as HIV education and treatment. The counseling program's theoretical orientation is described as client-centered.
- TAU Plus Galantamine (Experimental): Standard treatment plus Galantamine. In this study, we will use 8 mg galantamine extended release (ER). Galantamine ER is used once daily. The recommended initial dose is 8 mg/day and the maintenance dose is 16-24 mg/day.
  Interventions: Drug: Galantamine
- TAU plus Computer Assisted Cognitive Behavioral Therapy (CBT) (Experimental): TAU plus computer assisted CBT plus placebo. All participants assigned to this condition will also be offered up to 60 minutes per week to work with the CBT for CBT program, onsite at the clinic, in a private space and using a computer provided by the research project. Patients will have the choice of how they choose to use the computer, that is, in two 30-minute sessions or one one-hour session.
  Interventions: Behavioral: Computer Assisted Cognitive Behavioral Therapy (CBT)
- TAU plus CBT plus galantamine (Experimental): Standard treatment, plus computer assisted cognitive behavioral therapy, plus galantamine.
  Interventions: Drug: Galantamine; Behavioral: Computer Assisted Cognitive Behavioral Therapy (CBT)

INTERVENTIONS:
Drug: Galantamine — Daily 8 mg galantamine capsule
  Other Names: Nivalin, Razadyne, Razadyne ER, Reminyl, Lycoremine
  Arms: TAU Plus Galantamine; TAU plus CBT plus galantamine
Behavioral: Computer Assisted Cognitive Behavioral Therapy (CBT) — CBT a psychotherapeutic approach that addresses dysfunctional emotions, maladaptive behaviors and cognitive processes and contents through a number of goal-oriented, explicit systematic procedures. The name refers to behavior therapy, cognitive therapy, and to therapy based upon a combination of basic behavioral and cognitive principles and research.
  Arms: TAU plus CBT plus galantamine; TAU plus Computer Assisted Cognitive Behavioral Therapy (CBT)

SUMMARY:
We are testing to see if Galantamine, a learning enhancing medication, will help methadone maintained cocaine abusers with their learning and memory specific to CBT using an innovative CBT computer program.

DETAILED DESCRIPTION:
We are proposing a randomized double blind clinical trial of galantamine and our innovative computer-assisted version of CBT, alone and in combination, to improve treatment outcome and cognitive functioning among cocaine users. The proposed study will be the first to evaluate a cognitive enhancing medication as a means of enhancing the effects of an extremely promising empirically validated behavioral therapy for addiction, and hence bridge cognitive neuroscience and behavioral therapies development.

The aim is to conduct a 12 week randomized placebo controlled trial, using a 2x2 factorial model, that will evaluate the efficacy of adding computer assisted training in CBT ("CBT4CBT") and galantamine to standard treatment for 160 cocaine abusing or dependent methadone-maintained individuals. Participants will be randomized to (1) standard treatment (TAU) plus placebo, (2) TAU plus galantamine, (3) TAU plus CBT4CBT plus placebo, or (4) TAU plus CBT4CBT plus galantamine.

ELIGIBILITY:
Inclusion Criteria:

* Males and females between ages of 18 and 50
* Enrolled in RNP methadone program and stable on methadone for at least 3 weeks
* Current cocaine abuse or dependence according to DSM-IV criteria
* No current medical problems and normal ECG
* If female, not currently pregnant or breast feeding and using reliable birth control
* Fluent in English and have at least a 6th grade reading level
* Can commit to 12 weeks of treatment and are willing to be randomized

Exclusion Criteria:

* Current major psychiatric illness including mood, psychotic or anxiety disorder
* History of major medical illnesses including asthma, chronic obstructive lung disease, gastrointestinal ulcer, hepatic or renal impairment, cardiac rhythm disturbances
* Use of medications including beta blockers and NASAIDs
* Known allergy to Galantamine

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2007-12; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen M Carroll, Ph.D., Principal Investigator — Yale University
Locations (2):
- United States (2):
  - Kinsella Treatment Center (KTC), Bridgeport, Connecticut
  - Regional Network of Programs, Stratford, Connecticut

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be available to other researchers upon request. Please contact Dr. Carroll

REFERENCES:
- [Derived] Carroll KM, Nich C, DeVito EE, Shi JM, Sofuoglu M. Galantamine and Computerized Cognitive Behavioral Therapy for Cocaine Dependence: A Randomized Clinical Trial. J Clin Psychiatry. 2018 Jan/Feb;79(1):17m11669. doi: 10.4088/JCP.17m11669. PMID 29286595

RESULTS

PARTICIPANT FLOW:
Groups:
- Galantamine and CBT: Drug: Galantamine Daily 8 mg galantamine capsule
  Other Names:
  Nivalin, Razadyne, Razadyne ER, Reminyl, Lycoremine Behavioral: Computer Assisted Cognitive Behavioral Therapy (CBT) CBT a psychotherapeutic approach that addresses dysfunctional emotions, maladaptive behaviors and cognitive processes and contents through a number of goal-oriented, explicit systematic procedures. The name refers to behavior therapy, cognitive therapy, and to therapy based upon a combination of basic behavioral and cognitive principles and research.
- Galantamine Only: Drug: Galantamine Daily 8 mg galantamine capsule
  Other Names:
  Nivalin, Razadyne, Razadyne ER, Reminyl, Lycoremine
- Placebo and CBT: TAU plus computer assisted CBT plus placebo. All participants assigned to this condition will also be offered up to 60 minutes per week to work with the CBT for CBT program, onsite at the clinic, in a private space and using a computer provided by the research project. Patients will have the choice of how they choose to use the computer, that is, in two 30-minute sessions or one one-hour session.
- Placebo Only: Standard Treatment plus placebo for cocaine abusing or dependent methadone-maintained individuals. This consists of daily methadone visits plus one individual and one group session per week, and patients may participate in additional treatments such as HIV education and treatment. The counseling program's theoretical orientation is described as client-centered.
Period: Overall Study
Arm/Group | Galantamine and CBT | Galantamine Only | Placebo and CBT | Placebo Only
Started | 28 | 27 | 38 | 27
Completed | 20 | 20 | 27 | 25
Not Completed | 8 | 7 | 11 | 2
Not completed — Lost to Follow-up | 7 | 6 | 10 | 2
Not completed — Withdrawal by Subject | 1 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Galantamine: Drug: Galantamine Daily 8 mg galantamine capsule
  Other Names:
  Nivalin, Razadyne, Razadyne ER, Reminyl, Lycoremine
- Placebo and CBT: Computer assisted CBT plus placebo. All participants assigned to this condition will also be offered up to 60 minutes per week to work with the CBT for CBT program, onsite at the clinic, in a private space and using a computer provided by the research project. Patients will have the choice of how they choose to use the computer, that is, in two 30-minute sessions or one one-hour session.
- Total: Total of all reporting groups
Arm/Group | Galantamine and CBT | Galantamine | Placebo and CBT | Placebo Only | Total
Number analyzed (Participants) | 28 | 27 | 38 | 27 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.04 (8.72) | 38.70 (10.79) | 39.82 (8.99) | 36.30 (9.41) | 38.36 (9.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 15 | 19 | 16 | 62
  Male | 16 | 12 | 19 | 11 | 58
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 12 | 15 | 19 | 16 | 62
  African-American | 7 | 6 | 9 | 3 | 25
  Hispanic | 9 | 6 | 9 | 8 | 32
  Multiracial/Other | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Cocaine Use
Description: Reduction in cocaine use, operationalized as the frequency of cocaine use by month using timeline followback.
Time Frame: 12 weeks
Population: Presented are data for those measured at baseline and at 12 weeks. 2 individuals in the Galantamine arm were not measured at 12 weeks.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Galantamine and CBT | Galantamine | Placebo and CBT | Placebo Only
Number analyzed (Participants) | 28 | 27 | 38 | 27
Days
  Baseline | 18.82 (8.68) | 14.81 (9.05) | 15.68 (7.78) | 14.85 (8.47)
  12 Weeks: number analyzed (Participants) | 28 | 25 | 38 | 27
  12 Weeks | 8.60 (6.95) | 6.32 (6.52) | 7.65 (7.41) | 10.25 (7.79)

2. Primary Outcome: Cocaine Abstinence
Description: operationalized by percentage of drug-free urine specimens submitted (We will use the Branan ToxCup Drug Screen Cup onsite TESTCUP system for detection of cocaine, methamphetamine, THC, benzodiazepine, and opioids) at 12 Weeks
Time Frame: 12 weeks
Population: Three arm had one subject drop out before study medication was given- therefore the number analyzed are those that received first treatment.
Measure: Mean (Standard Deviation); unit: percentage of negative urines
Arm/Group | Galantamine and CBT | Galantamine | Placebo and CBT | Placebo Only
Number analyzed (Participants) | 27 | 26 | 37 | 27
percentage of negative urines | 22.45 (35.62) | 31.13 (34.16) | 20.49 (27.60) | 14.78 (19.11)

3. Secondary Outcome: Cognitive Function
Description: A composite using a carefully selected neuropsychological battery that includes measures of executive cognitive functioning frequently affected among cocaine users, likely to be important moderators of CBT4CBT, and sensitive to galantamine effects. These will include measures of multiple aspects of attention, cognitive inhibition, sustained attention (CANTAB), decision making (BART), and memory (digit span).
  Scores ranged from -1.77 to 1.42 with a higher score indicating higher cognitive functioning.
Time Frame: 12 weeks
Population: All participants did not complete the CANTAB assessments at both pre and post treatment. Reasons for not completing were refusal to complete the tasks, inability to complete the tasks in a manner in which they could be scored and equipment or computer problems.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Galantamine and CBT | Galantamine | Placebo and CBT | Placebo Only
Number analyzed (Participants) | 18 | 22 | 25 | 19
scores on a scale | -.12 (.58) | .11 (.50) | -.06 (.71) | .03 (.49)

ADVERSE EVENTS:
Arm/Group | Galantamine and CBT | Galantamine | Placebo and CBT | Placebo Only
Serious Adverse Events (participants affected / at risk) | 4/28 | 6/27 | 6/38 | 5/27
Other Adverse Events (participants affected / at risk) | 15/28 | 10/27 | 16/38 | 14/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Galantamine and CBT (N=28) | Galantamine (N=27) | Placebo and CBT (N=38) | Placebo Only (N=27)
Inpatient Substance Use Treatment Hospitalization (Psychiatric disorders) | 3 (5) | 2 (2) | 3 (5) | 5 (5)
Inpatient Psychiatric Hospitalization (Psychiatric disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Medical hospitalization (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Medical hospitalization (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Medical Hospitalization (General disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Galantamine and CBT (N=28) | Galantamine (N=27) | Placebo and CBT (N=38) | Placebo Only (N=27)
Fatigue (General disorders) | 2 (3) | 3 (5) | 8 (13) | 4 (7)
agitation (General disorders) | 4 (5) | 0 (0) | 3 (3) | 1 (1)
headache (General disorders) | 5 (6) | 6 (8) | 6 (9) | 3 (5)
Tremors (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dizziness (General disorders) | 3 (5) | 2 (3) | 2 (3) | 1 (1)
Nausea (Gastrointestinal disorders) | 11 (17) | 2 (2) | 5 (14) | 6 (6)
indigestion (Gastrointestinal disorders) | 2 (3) | 0 (0) | 3 (4) | 2 (2)
Blood in Stool (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal Pain (General disorders) | 4 (5) | 1 (1) | 4 (5) | 1 (1)
Loss of Appetite (General disorders) | 7 (10) | 2 (3) | 6 (8) | 3 (3)
Diarrhea or Constipation (Gastrointestinal disorders) | 4 (7) | 0 (0) | 8 (13) | 3 (3)
Weight Loss (General disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes